CLINICAL TRIAL: NCT03589391
Title: A New Pressure Guided Mechatronic Tool for Epidural Space Detection: Feasibility Assessment in a Clinical Scenario
Brief Title: New Mechatronic Device for Epidural Space Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Massimiliano Carassiti, Associate Professor, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Device Feasibility
Other Study IDs: EPISENS
Record Dates: First submitted 2018-07-06; First posted 2018-07-17 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Non Invasive Monitoring of Loss of Resistance During Epidural Injection
Keywords: Epidural injection; loss of resistance detection; mechatronic device

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Procedures with the use of device for LOR monitoring (Experimental): Patients enrolled suffered from chronic back pain and underwent epidural infiltration. The device is used.
  Interventions: Device: LOR measurement via device
- Procedures without the use of device for LOR monitoring (No Intervention): Patients enrolled suffered from chronic back pain and underwent epidural infiltration

INTERVENTIONS:
Device: LOR measurement via device — The epidural technique is totally performed in a sterile field without any harm to the patient. The LOR measurement is monitored via the bespoke device used during the epidural procedure.
  Arms: Procedures with the use of device for LOR monitoring

SUMMARY:
This study sought to perform the feasibility assessment of a new, non-invasive device for Loss of Resistance (LOR) detection in clinical settings. The device in charge is a mechatronic device optimized in its configurations in order to detect Loss of Resistance while performing epidural injections.

ELIGIBILITY:
Inclusion Criteria:

* patients whose pathology requires specific treatment such as epidural infiltration

Exclusion Criteria:

* coagulation abnormalities or assumption of anticoagulant drugs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-12-23 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
Loss of resistance detection | throughout the epidural infiltration procedure
  A non invasive device to detect loss of resistance during epidural infiltration

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Carassiti, MD, Principal Investigator — University Campus Bio-Medico of Rome
Locations (2):
- Italy (2):
  - Campus Bio Medico, Rome, RM
  - University Hospital Campus BioMedico, Rome

REFERENCES:
- [Background] Tesei M, Saccomandi P, Massaroni C, Quarta R, Carassiti M, Schena E, Setola R. A cost-effective, non-invasive system for pressure monitoring during epidural needle insertion: Design, development and bench tests. Annu Int Conf IEEE Eng Med Biol Soc. 2016 Aug;2016:194-197. doi: 10.1109/EMBC.2016.7590673. PMID 28268312
- [Background] Carassiti M, Biselli V, Cecchini S, Zanzonico R, Schena E, Silvestri S, Cataldo R. Force and pressure distribution using Macintosh and GlideScope laryngoscopes in normal airway: an in vivo study. Minerva Anestesiol. 2013 May;79(5):515-24. Epub 2013 Feb 18. PMID 23419341
- [Background] Carassiti M, Mattei A, Pizzo CM, Vallone N, Saccomandi P, Schena E. Bronchial blockers under pressure: in vitro model and ex vivo model. Br J Anaesth. 2016 Sep;117 Suppl 1:i92-i96. doi: 10.1093/bja/aew120. Epub 2016 Jun 14. PMID 27307290
- [Background] Carassiti M, Mattei A, Quarta R, Massaroni C, Saccomandi P, Tesei M, Setola R, Schena E. A New Pressure Guided Management Tool for Epidural Space Detection: Feasibility Assessment on a Simulator. Artif Organs. 2017 Dec;41(12):E320-E325. doi: 10.1111/aor.13007. Epub 2017 Oct 25. PMID 29068081
- [Background] Carassiti M, Quarta R, Mattei A, Tesei M, Saccomandi P, Massaroni C, Setola R, Schena E. Ex vivo animal-model assessment of a non-invasive system for loss of resistance detection during epidural blockade. Annu Int Conf IEEE Eng Med Biol Soc. 2017 Jul;2017:759-762. doi: 10.1109/EMBC.2017.8036935. PMID 29059983